CLINICAL TRIAL: NCT00835510
Title: A Randomized, Double-Blind, Placebo Controlled, Parallel Design, Multiple-Site Study to Evaluate the Clinical Equivalence of Two Butenafine Hydrochloride 1% Creams in Patients With Interdigital Tinea Pedis
Brief Title: Clinical Equivalence of Two Butenafine Hydrochloride 1% Creams in Patients With Interdigital Tinea Pedis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BTNF-0708
Record Dates: First submitted 2009-01-30; First posted 2009-02-03 (Estimated); Results first posted 2009-10-06 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-01

CONDITIONS: Tinea Pedis
Keywords: Tinea pedis
MeSH Terms: conditions — Tinea Pedis | interventions — butenafine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Butenafine cream 1% (Taro) (Experimental): Butenafine cream manufactured by Taro applied for 7 days
  Interventions: Drug: Butenafine cream 1% manufactured by Taro
- Lotrimin Ultra (butenafine) 1% (Active Comparator): Lotrimin Ultra (butenafine) applied for 7 days
  Interventions: Drug: Lotrimin Ultra (butenafine) 1%
- Vehicle (Placebo Comparator): Butenafine vehicle applied for 7 days
  Interventions: Drug: Butenafine Vehicle manufactured by Taro

INTERVENTIONS:
Drug: Butenafine cream 1% manufactured by Taro — Treatment applied to affected area twice daily for 7 days
  Arms: Butenafine cream 1% (Taro)
Drug: Lotrimin Ultra (butenafine) 1% — Treatment applied to affected area twice daily for 7 days
  Arms: Lotrimin Ultra (butenafine) 1%
Drug: Butenafine Vehicle manufactured by Taro — Treatment applied to affected area twice daily for 7 days
  Arms: Vehicle

SUMMARY:
To demonstrate comparable safety and efficacy of Taro Pharmaceuticals Inc. butenafine hydrochloride cream 1% (test product) and Lotrimin Ultra® cream (reference listed drug) in the treatment of interdigital tinea pedis, and to show the superiority of the active treatments over that of the placebo (vehicle).

ELIGIBILITY:
Inclusion Criteria:

* Microbiologically confirmed clinical diagnosis of interdigital tinea pedis
* If female and of child bearing potential, prepare to abstain from sexual intercourse or use a reliable method of contraception during the study (e.g., condom, intra-uterine device (IUD), oral, transdermal, injected or implanted hormonal contraceptives).
* A confirmed clinical diagnosis of interdigital tinea pedis. Lesions are to be predominately interdigital but may extend to other areas of the foot (the non-interdigital lesions must not be hyperkeratotic).
* The presence of tinea pedis infection, confirmed by the observation of segmented fungal hyphae during a microscopic potassium hydroxide (KOH) wet mount examination (potassium hydroxide mount preparation).
* Identification of an appropriate dermatophyte by culture sent to the central laboratory. The appropriate dermatophytes are Trichophyton rubrum, Trichophyton mentagrophyte or Epidermophyton floccosum.

Exclusion Criteria:

* Use of any of the following within the indicated timeline:
* Oral or injectable steroids
* Any oral anti-fungals within 4 weeks of the study start
* Use of topical corticosteroids or any other topical antipruritics on the feet within 72 hours of the study start.
* Any prescription or over-the-counter (OTC) topical antifungals on the feet within two weeks prior to study entry
* Use of any antihistamines within 72 hours of the study start.
* Any known hypersensitivity to butenafine or other antifungal agents.
* Evidence of any concurrent dermatophytic infection of toe nails (onychomycosis) or other dermatological condition of the foot that may interfere with the Investigator's evaluation of tinea pedis.
* Patients with recurrent tinea pedis (more than 3 infections in the past 12 months) who have been unresponsive to previous antifungal therapy.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 548 (Actual)
Dates: Start 2008-06; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (16):
  - Investigator Site, Burbank, California
  - Investigator Site, San Diego, California
  - Investigator Site, Miami, Florida
  - Investigator Site, Martinez, Georgia
  - Investigator Site, Stockbridge, Georgia
  - Investigator Site, Clinton Township, Michigan
  - Investigator Site, Hickory, North Carolina
  - Investigator Site, Raleigh, North Carolina
  - Investigator Site, Salisbury, North Carolina
  - Investigator Site, Sylvania, Ohio
  - Investigator Site, Simpsonville, South Carolina
  - Investigator Site, Bristol, Tennessee
  - Investigator Site, Nashville, Tennessee
  - Investigator Site, College Station, Texas
  - Investigator Site, Houston, Texas
  - Investigator Site, San Antonio, Texas
- Investigator Site, Belize City, Belize

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients 12 years of age and older, who presented with interdigital tinea pedis, with a positive potassium hydroxide test (KOH) and met the inclusion/exclusion criteria were enrolled in the trial. Subsequently samples were sent for culture to confirm that either T. rubrum, T. mentagrophytes, or E. floccosum were the causative organism.
Period: Overall Study
Arm/Group | Butenafine Cream 1% (Taro) | Lotrimin Ultra (Butenafine) 1% | Vehicle
Started | 219 | 221 | 108
Positive Fungal Culture | 149 | 155 | 71
Completed | 143 | 152 | 70
Not Completed | 76 | 69 | 38

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Butenafine Cream 1% (Taro) | Lotrimin Ultra (Butenafine) 1% | Vehicle | Total
Number analyzed (Participants) | 149 | 155 | 71 | 375
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 6 | 2 | 12
  Between 18 and 65 years | 135 | 142 | 66 | 343
  >=65 years | 10 | 7 | 3 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 41 | 23 | 106
  Male | 107 | 114 | 48 | 269
Region of Enrollment [Number; unit: participants]
  United States | 123 | 135 | 62 | 320
  Belize | 26 | 20 | 9 | 55

OUTCOME MEASURES:

1. Primary Outcome: Therapeutic Cure - Superiority Analysis
Description: Therapeutic Cure requires both Clinical Cure and Mycological Cure.
  Clinical Cure was based on the following signs and symptoms: fissuring, erythema, maceration, vesiculation, scaling, exudation, pruritus, burning. Each clinical symptom was evaluated using a 0-3 point rating scale: none=0, mild=1, moderate=2 or severe=3. If the score for erythema was ≤ 2 and the sum for all of the other 7 signs and symptoms was <2 then the patient was considered a Clinical Cure.
  Mycological Cure: The potassium hydroxide (KOH) and the fungal culture were both negative.
Time Frame: 42 days
Population: Patients with negative cultures at baseline are excluded. Efficacy ITT analysis includes all patients with positive baseline cultures, who received at least one dose of medication, had a follow-up visit and had data for the day 42 visit.
Measure: Number; unit: Participants
Arm/Group | Butenafine Cream 1% (Taro) | Lotrimin Ultra (Butenafine) 1% | Vehicle
Number analyzed (Participants) | 143 | 152 | 70
Participants | 76 | 108 | 24
Statistical Analysis 1: Comparison: Butenafine Cream 1% (Taro) vs Vehicle; Test type: Superiority or Other; p = 0.0127, Fisher Exact; two-sided
Statistical Analysis 2: Comparison: Lotrimin Ultra (Butenafine) 1% vs Vehicle; Test type: Superiority or Other; p < 0.0001, Fisher Exact; two-sided

2. Secondary Outcome: Therapeutic Cure
Description: Subject with clinical and mycological cure at day 7
Time Frame: 7 days
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Butenafine Cream 1% (Taro) | Lotrimin Ultra (Butenafine) 1% | Vehicle
Number analyzed (Participants) | 149 | 153 | 71
Participants | 30 | 38 | 11

3. Secondary Outcome: Mycologic Cure
Description: Negative KOH and fungal culture at day 42
Time Frame: 42 days
Population: ITT population
Measure: Number; unit: Participants
Arm/Group | Butenafine Cream 1% (Taro) | Lotrimin Ultra (Butenafine) 1% | Vehicle
Number analyzed (Participants) | 141 | 152 | 70
Participants | 101 | 128 | 33

4. Secondary Outcome: Clinical Cure
Description: The following 8 signs and symptoms are rated at each visit:
  Erythema Fissuring Maceration Vesiculation Desquamation/scaling Exudation Pruritus Stinging/Burning
  Each symptom is evaluated using the following scale:
  0 = None- Complete absence of any sign or symptom
  1. = Mild - obvious but minimal involvement
  2. = Moderate - something that is easily noted
  3. = Severe - quite marked
  Clinical cure is defined as a score of 2 (moderate) or less for erythema and a total score for seven other signs and symptoms less than 2.
Time Frame: 42 days
Population: ITT population
Measure: Number; unit: Participants
Arm/Group | Butenafine Cream 1% (Taro) | Lotrimin Ultra (Butenafine) 1% | Vehicle
Number analyzed (Participants) | 142 | 152 | 70
Participants | 83 | 111 | 27

5. Secondary Outcome: Safety and Adverse Event Profile
Time Frame: 42 days
Reporting Status: Not Posted

6. Primary Outcome: Therapeutic Cure Non-Inferiority Comparison of Butenafine Cream and Lotrimin Ultra
Description: Patient was cured both by symptoms (Clinical Cure) and by the results of fungal testing (Mycological Cure).
Time Frame: 42 days
Population: Patients with negative cultures excluded. Use per protocol population
Measure: Number; unit: Participants
Arm/Group | Butenafine Cream 1% (Taro) | Lotrimin Ultra (Butenafine) 1% | Vehicle
Number analyzed (Participants) | 126 | 139 | 0
Participants | 63 | 97 |
Statistical Analysis 1: Comparison: Butenafine Cream 1% (Taro) vs Lotrimin Ultra (Butenafine) 1%; Test type: Non-Inferiority or Equivalence — The criteria for equivalence is that the 90% confidence interval for the difference in cure rate had to be between -20% to +20%; Cure rate difference = -19.78, 90% CI [-30.27 to -9.29]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the 42 day duration of the study.
Description: The Safety Population includes all 548 patients who received at least a single dose of medication.
Arm/Group | Butenafine Cream 1% (Taro) | Lotrimin Ultra (Butenafine) 1% | Vehicle
Serious Adverse Events (participants affected / at risk) | 2 | 0 | 1
Other Adverse Events (participants affected / at risk) | 14 | 21 | 5
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Butenafine Cream 1% (Taro) | Lotrimin Ultra (Butenafine) 1% | Vehicle
Cellulitis (Infections and infestations) | 1/219 (1) | 0/221 (0) | 1/108 (1)
Tachycardia (Cardiac disorders) | 1/219 (1) | 0/221 (0) | 0/108 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Butenafine Cream 1% (Taro) | Lotrimin Ultra (Butenafine) 1% | Vehicle
Headache (Nervous system disorders) | 10/219 (10) | 16/221 (16) | 4/108 (4)
Nasopharyngitis (Infections and infestations) | 4/219 (4) | 5/221 (5) | 1/108 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days